CLINICAL TRIAL: NCT06476548
Title: Mindfulness-Based Ecological Momentary Intervention For Smoking Cessation Among Cancer Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MCC-22266; K99CA271040 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Any Cancer Type
Keywords: Smoking Cessation; Cancer Survivor
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usability Testing (Experimental): Participants will receive brief counseling, nicotine replacement therapy, and intervention content delivered via the app.
  Interventions: Device: EMI

INTERVENTIONS:
Device: EMI — Participants will complete 3 counseling sessions (30 minutes), download and use a smartphone app for 4 weeks, complete 2 online surveys, and a brief phone call at the end of the study to provide feedback. In the first 3 weeks, participants will use the prototype app every day to complete ecological momentary assessments (EMAs), receive brief mindful skills, and practice formal mindfulness meditations (5-20 minutes). In the final week, participants will continue completing EMAs. Participants will also be provided with nicotine patches.

SUMMARY:
The purpose of the study is to obtain feedback on a new quit-smoking treatment among individuals with a cancer diagnosis using a prototype app we developed.

DETAILED DESCRIPTION:
The study aims to test the usability of the prototype app in conjunction with face-to-face brief cessation counseling and nicotine replacement therapy in a single-arm trial.

ELIGIBILITY:
Inclusion Criteria:

* Having smoked at least one cigarette (even one or two puffs) within the past 30 days.
* Having been diagnosed with cancer.
* Willing to give quitting a try as part of the study.
* Having a smartphone that allows installation of the app.
* Willingness to download and use the app daily.
* Valid home address and functioning phone number.
* Being able to read, write, and speak English.

Exclusion Criteria:

* Being enrolled in a smoking cessation program.
* Current use of smoking cessation medications.
* Evidence of current psychosis.
* Current/planning pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, PhD, Principal Investigator — Moffitt Cancer Center; Min-Jeong Yang, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usability Testing
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Usability Testing
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 0
  40-49 | 3
  50-59 | 3
  60-69 | 6
  70-79 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Percentage of participants who downloaded the study's smartphone application and attended the first counseling session.
Time Frame: At 4 weeks
Measure: Number; unit: percentage of Participants
Arm/Group | Usability Testing
Number analyzed (Participants) | 12
percentage of Participants | 91.7

2. Primary Outcome: Likability of Mindfulness Practices
Description: Participants will rate the likability of mindfulness practices delivered through the study app on a 6-point Likert scale from 1 (Extremely dislike) to 6 (Extremely like).
Time Frame: At 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Usability Testing
Number analyzed (Participants) | 11
score on a scale | 6 [2 to 6]

3. Primary Outcome: Utility of Mindfulness Practices
Description: Participants will rate their perceived helpfulness of mindfulness practices delivered through the study app on a 6-point Likert scale from 1 (Extremely unhelpful) to 6 (Extremely helpful).
Time Frame: At 4 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Usability Testing
Number analyzed (Participants) | 11
score on a scale | 5 [1 to 6]

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Usability Testing
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT06476548/Prot_SAP_000.pdf